CLINICAL TRIAL: NCT00183326
Title: Treating PTSD in Children Exposed to Domestic Violence
Brief Title: Treating Post Traumatic Stress Disorder in Children Exposed to Domestic Violence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Judith Cohen, Physician, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH072590 (NIH); R01MH072590 (NIH); DDTR B3-PDS
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Stress Disorders, Post-Traumatic; Anxiety; Depression
Keywords: Posttraumatic Stress Disorder; Domestic Violence; Children; Cognitive Behavioral Therapy; CBT
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive trauma-focused cognitive behavioral therapy
  Interventions: Behavioral: Trauma-focused cognitive behavioral therapy (TF-CBT)
- 2 (Active Comparator): Participants will receive child-centered supportive therapy
  Interventions: Behavioral: Child-centered supportive therapy (CCT)

INTERVENTIONS:
Behavioral: Trauma-focused cognitive behavioral therapy (TF-CBT) — TF-CBT is a psychotherapeutic intervention designed to help children, youth, and their parents overcome the negative effects of traumatic life events. It was developed by integrating cognitive and behavioral interventions with traditional child abuse therapies that focus on enhancement of interpersonal trust and empowerment. It targets PTSD symptoms, which often co-occur with depression and behavioral problems. TF-CBT also targets other issues experienced by those suffering a trauma including poor self-esteem, mood instability, and difficulty trusting others.
  Arms: 1
Behavioral: Child-centered supportive therapy (CCT) — CCT demonstrates an empathic approach to healing. An environment consisting of empathy, unconditional positive regard and acceptance are key elements in this mode of therapy.
  Arms: 2

SUMMARY:
This study will determine whether trauma-focused cognitive behavioral therapy (TF-CBT) is more effective than child-centered therapy (CCT) in reducing post traumatic stress disorder (PTSD) in children exposed to domestic violence (DV).

DETAILED DESCRIPTION:
Up to 10 million children in the United States are exposed to DV directed at their mothers by intimate partners. DV exposure puts these children at an increased risk for developing behavioral problems, depression, anxiety, and PTSD. While studies targeting PTSD in DV-exposed children are limited, data indicates that TF-CBT is effective in improving PTSD as well as depression, anxiety, and behavioral symptoms. This study will determine the effectiveness of TF-CBT in reducing PTSD and other DV-related psychological symptoms in children from a community DV agency in Pittsburgh, Pennsylvania.

This study will last 8 weeks. Children and their mothers will be randomly assigned to receive 8 weeks of either TF-CBT or CCT. In TF-CBT, patients recall the events of their trauma and try to deal with the emotions that arise. Supportive treatment empowers children to deal with their emotions in general. Both the children and their mothers will complete questionnaires at study entry and at Week 8. Children will also complete self-report scales at study entry and at Week 8. The questionnaires and self-report scales will be used to assess symptoms of PTSD, depression, anxiety, and behavioral problems. Children and their mothers will be contacted 6 and 12 months after study completion for follow-up interviews.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PTSD related to exposure to DV, defined as their mother having been the victim of intimate partner violence within 1 year prior to study entry
* Able to read and understand English
* Parent or guardian able to read and understand English
* Parent or guardian willing to give informed consent

Exclusion Criteria:

* Certain psychiatric disorders which preclude participation in cognitive-based treatment

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 124 (Actual)
Dates: Start 2004-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
PTSD symptoms | Measured before and after treatment and Months 6 and 12 of follow-up
Anxiety | Measured before and after treatment and Months 6 and 12 of follow-up
Depression | Measured before and after treatment and Months 6 and 12 of follow-up
Behavior | Measured before and after treatment and Months 6 and 12 of follow-up

SECONDARY OUTCOMES:
Contact with perpetrator | Measured at every treatment session

CONTACTS AND LOCATIONS:
Overall Officials: Judith A. Cohen, MD, Principal Investigator — Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Locations (1):
- Women's Center and Shelter of Greater Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Cohen JA, Mannarino AP, Iyengar S. Community treatment of posttraumatic stress disorder for children exposed to intimate partner violence: a randomized controlled trial. Arch Pediatr Adolesc Med. 2011 Jan;165(1):16-21. doi: 10.1001/archpediatrics.2010.247. PMID 21199975
- See also: Click here to learn more about the National Child Traumatic Stress Network — https://www.nctsn.org